CLINICAL TRIAL: NCT06172621
Title: Spinal Cord Associative Plasticity for Amyotrophic Lateral Sclerosis
Brief Title: Spinal Cord Associative Plasticity for ALS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: B4258-R; 1I01RX004258 (NIH)
Record Dates: First submitted 2023-12-06; First posted 2023-12-15 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: neuromodulation; spinal cord stimulation; task-oriented exercise; transcranial magnetic stimulation
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: After a run-in phase of 2-4 months to determine individualized stimulation parameters, participants will be randomized into Group A and Group B. Group A will undergo 2 weeks (6 sessions) of SCAP alone. Group B will undergo 2 weeks (6 sessions) of SCAP plus upper extremity task-oriented exercise.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SCAP alone (Active Comparator): After a run-in phase of 2-4 months to determine individualized stimulation parameters, participants will be randomized into a comparator group of two weeks (6 sessions) of SCAP intervention alone.
  Interventions: Procedure: Spinal Cord Associative Plasticity (SCAP)
- SCAP plus task-oriented exercise (Experimental): After a run-in phase of 2-4 months to determine individualized stimulation parameters, participants will be randomized into a comparator group of two weeks (6 sessions) of SCAP intervention plus upper extremity task-oriented exercise.
  Interventions: Procedure: Spinal Cord Associative Plasticity (SCAP); Procedure: Upper extremity task-oriented exercise

INTERVENTIONS:
Procedure: Spinal Cord Associative Plasticity (SCAP) — Paired non-invasive brain and spinal cord stimulation.
Procedure: Upper extremity task-oriented exercise — Participants will perform a range of exercises composed of tasks resembling daily home/community activities such as stacking and sorting small objects, manipulating writing utensils, keys, buttons, etc.
  Arms: SCAP plus task-oriented exercise

SUMMARY:
Veterans are at higher risk than non-Veterans of falling ill with amyotrophic lateral sclerosis (ALS).

The investigators have shown that synchronized stimulation over the brain and cervical spinal cord can temporarily strengthen weakened nerve circuits between the brain and hand muscles in people with ALS.

The current proposal will take the next step of individualizing this intervention, then applying it repetitively in an attempt to achieve direct clinical benefit on hand strength and function.

Following an initial 2-3 month period of optimizing the intervention for each individual, the investigators will compare the effects of two-week programs of paired brain-spinal stimulation with or without hand exercises.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is more prevalent in Veterans than civilians, leading to ALS being considered a Service-Connected condition by the VA. ALS features incomplete degeneration of upper and lower motor neuron pathways within the spinal cord, a circumstance resembling that of spinal cord injury (SCI). Transcutaneous spinal cord stimulation (TSCS) has demonstrated remarkable potential to activate damaged circuits after SCI to improve motor and autonomic function.

Partly funded by a prior VA award (RX002527), the investigators have preliminary data demonstrating that pairing subthreshold cervical TSCS pulses with suprathreshold transcranial magnetic stimulation (TMS) pulses can enhance hand muscle motor evoked potentials when the cortical pulse reaches the cervical spinal cord 0-5 milliseconds prior to the spinal pulse. This evidence for immediate facilitation of the response to one pair of pulses suggests that if given repetitively, this approach could mediate spinal cord associative plasticity (SCAP) outlasting the period of paired stimulation. The investigators propose that increasing neural plasticity in this manner could be applied as a method to strengthen volitional (cortical) motor output and/or to 'prime' weakened circuits for improved responses to task-oriented exercise.

Both exercise and neuromodulation are understudied in ALS. Though not likely to cure the underlying disease mechanism, these approaches have the potential to mediate symptomatic benefit. The investigators strive to find better ways to conduct disease-oriented research that may provide direct clinical benefit to research participants with ALS and simultaneously increase scientific understanding. Additionally, most ALS clinical study entry criteria heavily favor those at earlier stages of disease. Strict entry criteria are understandable from the scientific perspective. However, we have repeatedly observed the frustration and rejection felt by individuals with ALS who cannot enter clinical trials. This proposed study does not restrict entry by time since symptom onset. The investigators thereby hope to produce more generalizable knowledge by performing a phased study:

1. Optimization: SCAP synaptic pairing interval and repetitive frequency pattern will be individually optimized to enhance hand muscle excitability and dexterity. The investigators hypothesize that pairs of stimuli with TMS arriving at the cervical spinal cord up to 2 ms prior to TSCS, delivered in an 'intermittent theta burst' pattern, will produce the strongest facilitation of hand neural circuits.
2. Consolidation: Two-week programs of SCAP alone versus SCAP plus task-oriented hand exercise will be compared. The investigators hypothesize that the combined intervention will result in greater and longer lasting physiological and clinical benefits than SCAP by itself.

There are currently no clinical studies in the world involving magnetic brain paired with phasic electrical spinal stimulation for ALS. Therefore, safety needs to be meticulously tracked. Aside from detailed clinical safety measures, the investigators will analyze serum biomarkers drawn at baseline and various stages of the study to better understand whether baseline levels of neurodegenerative, excitotoxic, inflammatory, and neurotropic biomarkers associate with either beneficial or detrimental responses to SCAP and exercise interventions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ALS by Gold Coast Criteria (Shefner et al. 2020) or "definite" or "probable" ALS by revised El Escorial Criteria (Brooks et al. 2000)
* Incomplete weakness: Score of 1, 2, 3, or 4 (out of 5) on manual muscle testing of finger extension, finger flexion, or finger abduction in left or right hand
* TSCS-evoked potential amplitude of at least 25 V in left or right abductor pollicis brevis (APB) or first dorsal interosseous (FDI) muscles with a resting motor threshold of 55 mA or lower
* TMS-evoked potential amplitude of at least 25 V in left or right abductor pollicis brevis (APB) or first dorsal interosseous (FDI) muscles with a resting motor threshold of 65% MSO or lower

Exclusion Criteria:

* History of seizures
* Ventilator dependence or patent tracheostomy site
* Use of medications that significantly lower seizure threshold, such as amphetamines and dalfampridine
* History of severe head trauma (evidence of brain contusion or hemorrhage or depressed skull fracture on prior imaging)
* History of implanted brain/spine/nerve stimulators, aneurysm clips, ferromagnetic metallic implants in the head (except for inside mouth); cochlear implants; cardiac pacemaker/defibrillator; intracardiac lines; currently increased intracranial pressure; or other contraindications to brain or spine stimulation
* Significant coronary artery or cardiac conduction disease; heart failure with an ejection fraction of less than 30% or with a New York Heart Association Functional Classification of Class III or IV
* History of significant tinnitus
* History of bipolar disorder
* History of suicide attempt
* Active psychosis
* Ongoing illicit drug or alcohol abuse in the past 6 months
* Heavy alcohol consumption (greater than equivalent of 5 ounces of liquor) within previous 48 hours
* Open skin lesions over the neck, shoulders, or arm stimulation or recording sites
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Amplitude of intrinsic hand muscle response to single-pulse transcranial magnetic stimulation (TMS) | Through study completion, up to 6 months
  The primary neurophysiological outcome will be corticospinal excitability measured at the first dorsal interosseous (FDI) muscle. If no suitable FDI muscle, will substitute with abductor pollicis brevis (APB) muscle.
Hand dexterity on the nine-hole peg test | Through study completion, up to 6 months
  Time to complete placement of nine pegs into their respective holes using the target hand.

SECONDARY OUTCOMES:
Volitional strength assessed by isometric dynamometry (key-pinch configuration) | Through study completion, up to 6 months
  Maximal isometric pinch strength will be measured using a pinch dynamometer. Maximum volitional force will be applied for 3-5 seconds, with at least 30 seconds between trials. The highest achieved value will be used for analysis.
Volitional strength assessed by isometric dynamometry (tip-to-tip configuration) | Through study completion, up to 6 months
  Maximal isometric pinch strength will be measured using a pinch dynamometer. Maximum volitional force will be applied for 3-5 seconds, with at least 30 seconds between trials. The highest achieved value will be used for analysis.
Volitional strength assessed by isometric dynamometry (grip configuration) | Through study completion, up to 6 months
  Maximal isometric pinch strength will be measured using a hand dynamometer. Maximum volitional force will be applied for 3-5 seconds, with at least 30 seconds between trials. The highest achieved value will be used for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Noam Y. Harel, MD PhD, Principal Investigator — James J. Peters Veterans Affairs Medical Center
Locations (1):
- James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified IPD will be deposited at Open Data Commons for Spinal Cord Injury
Supporting Information: Study Protocol, SAP
Time Frame: Within 1 year after study completion.
Access Criteria: Permanent
URL: https://odc-sci.org/